CLINICAL TRIAL: NCT01673425
Title: Evaluating Immune Response to Seasonal FluMist in Healthy Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual(4 completed subjects over 2 months)& inconclusive nasal wash assays.
Sponsor: National Center for Occupational Health and Infection Control (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB 604-2010
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2014-08

CONDITIONS: Influenza
Keywords: Influenza; Influenza Vaccines; Vaccines, Attenuated; Immunity, Mucosal
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Live Attenuated Influenza Vaccine (Experimental): Single intervention study- all participants will receive LAIV instead of injectable flu vaccine.
  Interventions: Drug: Live Attenuated Influenza Vaccine

INTERVENTIONS:
Drug: Live Attenuated Influenza Vaccine — All participants will be given FluMist.
  Other Names: FluMist

SUMMARY:
The Live-Attenuated Influenza Vaccine (LAIV), also known as FluMist, has been shown to be effective in children but less effective in adults. Our hypothesis is that this relative failure is due to adults having enough anti-flu IgA antibody in nasal secretions to neutralize the weakened vaccine virus.

DETAILED DESCRIPTION:
This is a VA-based study to evaluate serum and nasal wash antibody responses to seasonal LAIV of healthy Veterans and VA employees between the ages of 20 and 49 years old.

Specific Aims

1. The primary aim of the study is to evaluate whether people with high mucosal IgA antibodies against flu have a lower immune response to the seasonal LAIV.
2. The secondary objective is to determine whether the nasal wash viral neutralization data predicts LAIV immunization failures.

ELIGIBILITY:
Inclusion Criteria:

* Medically eligible healthy men and women between the ages of 20 to 49 years old.

Exclusion Criteria:

* A medical condition that places them at high risk for complications from influenza, including those with chronic heart or lung disease, such as asthma or reactive airway disease; people with medical conditions such as diabetes or kidney failure; or people with illnesses that weaken the immune system, or who take medications that can weaken the immune system.
* A history of Guillain-Barré Syndrome that occurred after receiving influenza vaccine
* Currently pregnant
* Have a severe allergy to chicken eggs or who are allergic to any of the nasal spray vaccine components
* Have had flu within the current flu season.
* Have had a flu vaccine within the current flu season.
* Have close contact with someone whose immune system is so weak they require care in a protected environment (such as bone marrow transplant unit).

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J. Radonovich, MD, Principal Investigator — National Center for Occupational Health and Infection Control
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Live Attenuated Influenza Vaccine: Single intervention study; all participants receive LAIV
Period: Overall Study
Arm/Group | Experimental: Live Attenuated Influenza Vaccine
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Live Attenuated Influenza Vaccine Study: This study was terminated due to poor enrollment and inconclusive nasal wash samples. No analyses were performed.
Arm/Group | Live Attenuated Influenza Vaccine Study
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: IgA Antibody Titers
Time Frame: Change from baseline in antibody titer at 6 weeks
Population: This study was terminated due to poor enrollment. Analyses were not conducted due to inconclusive nasal wash samples.
Groups:
- Experimental: Live Attenuated Influenza Vaccine: Single Intervention Study
Arm/Group | Experimental: Live Attenuated Influenza Vaccine
Number analyzed (Participants) | 0

2. Secondary Outcome: Serum Antibody Response to LAIV
Time Frame: Change from baseline in serum antibody response at 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Study Enrollment: Low accrual. Only 4 subjects completed study in 2 month period. Study terminated.
Arm/Group | Study Enrollment
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This study was terminated due to poor enrollment. Analyses were not conducted due to inconclusive nasal wash samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes